CLINICAL TRIAL: NCT06969976
Title: Effect of Immediate Use of Dry Cupping on Muscle Strength in Normal Adults
Brief Title: the Effect of Dry Cupping on Muscle Strength in Normal Individual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa S Ali, associate professor of pediatric physical therapy, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O6U.PT.REC/024/002001
Record Dates: First submitted 2025-05-02; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Normal Adults; Student Education
Keywords: adults; dry cupping; muscle strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): using dynamometer for the immediate effect of strengthening exercise for biceps muscle (biceps curl) without the application of dry cupping
  Interventions: Procedure: curl exericse
- experimental group (Experimental): using dynamometer for the immediate effect of strengthening exercise for biceps muscle during the application of dry cupping
  Interventions: Procedure: dry cupping and curl exercise

INTERVENTIONS:
Procedure: curl exericse — we use the curl exercise for control group to investigate the immediate effect of it on muscle strength in normal adults
  Other Names: curl exercise
  Arms: control group
Procedure: dry cupping and curl exercise — use dynamometer to measure biceps muscle strength in normal adults during the application of dry cupping with curl exercise
  Arms: experimental group

SUMMARY:
assessment of strengthening exercise during the application of dry cupping in normal adults

DETAILED DESCRIPTION:
this study will be conducted to answer the following questions: is the application of dry cupping will be effective during strengthening biceps muscle in normal adults who randomly assigned to 2 groups

ELIGIBILITY:
Inclusion Criteria:

* age ranges from 20 to 25 years
* the assessment is done on dominant hand

Exclusion Criteria:

* age >25 and <20 years
* having any problem in the tested upper limb (disease affecting shoulder, elbow, wrist and hand)
* having any cardiovascular problems
* cervical disorders affecting upper limb

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — to define muscle strength with error as there is difference between both gender in muscle strength
Enrollment: 84 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
strength of biceps muscle | Day 1
  use active force 2 dynamometer to measure the strength of biceps muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No